CLINICAL TRIAL: NCT00552331
Title: Prospective Randomized Clinical Study to Evaluate the Effects of Less Invasive Stabilization System (LISS) Plating Techniques in Distal Femoral Fractures
Brief Title: Evaluation of the Effects of Less Invasive Stabilization System (LISS) Plating Techniques in Distal Femoral Fractures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Synthes Canada (Industry); AO Research Fund (Other)
Responsible Party: Ross Leighton, MD, Capital District Health Authority, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDHA-RL-003
Record Dates: First submitted 2007-10-30; First posted 2007-11-01 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2009-05

CONDITIONS: Femoral Fractures
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LISS (Active Comparator): Treatment of distal femur fracture with less invasive stabilization system
  Interventions: Device: LISS
- Standard Treatment (Active Comparator): Treatment of distal femoral fractures using locking condylar plates or dynamic condylar screws
  Interventions: Device: Plates to treat fractures of the distal femur

INTERVENTIONS:
Device: Plates to treat fractures of the distal femur — use of dynamic condylar screws or locking condylar plates in the treatment of distal femur fractures
  Arms: Standard Treatment
Device: LISS — treatment of distal femur fractures with less invasive stabilization systems
  Arms: LISS

SUMMARY:
The purpose of this study is to determine whether the rate of fracture healing and fracture union, repaired with the LISS device, will be as good as or better than the usual fracture fixation systems.

ELIGIBILITY:
Inclusion Criteria:

* The patient has read and agree to the consent
* Patient is 16 years or older (bones have finished growing)
* The injury happened in the last 14 days

Exclusion Criteria:

* The patient taking part in another study
* The patient has an infection at the operative site
* The patient has a health condition that affects bone healing or interferes with their ability to complete the study requirements (questionnaires, examinations), for example Paget's disease or osteomalacia
* The patient is taking medication that affects bone healing (such as systemic steroids)
* The patient has malignant (tumor) disease
* The patient is unable to attend follow-up clinic visits

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2003-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Delayed union or nonunion of the distal femur | 12 months post operative
  Determined via radiographic analysis

SECONDARY OUTCOMES:
Time to clinical healing | 12 months
  assessed by weight-bearing ability and pain
Function as assessed by patient | 6 months, 12 months
  Assessed using LEM, SMFA, and SF-36 questionnaires
Frequency of adverse events | 12 months
Range of motion | Post-op, 6 weeks, 3 months, 6 months, 12 months
Gait analysis | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ross K Leighton, MD, FRCS(C), Principal Investigator — Capital Health, Canada
Locations (1):
- QEII Health Sciences Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Claireaux HA, Searle HKC, Parsons NR, Griffin XL. Interventions for treating fractures of the distal femur in adults. Cochrane Database Syst Rev. 2022 Oct 5;10(10):CD010606. doi: 10.1002/14651858.CD010606.pub3. PMID 36197809